CLINICAL TRIAL: NCT01394991
Title: A Randomized, Open-Label, Multicenter Study Evaluating Thrombovascular Events in Subjects With Cancer Receiving Chemotherapy and Administered Epoetin Alfa Once or Three Times a Week for the Treatment of Anemia
Brief Title: A Safety Study of Epoetin Alfa in Patients With Cancer Who Have Chemotherapy-Related Anemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Senior Director, CDTL PROCRIT/EPREX, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR010543; EPOANE4008
Record Dates: First submitted 2010-09-10; First posted 2011-07-15 (Estimated); Results first posted 2011-07-15 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Anemia; Neoplasms
Keywords: Epoetin alfa (EPREX, ERYPO)
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

ARMS (2):
- 001 (Experimental): Epoetin alfa 450 IU/kg once a week (QW) 450 IU/kg once a week (QW) by subcutaneous injection preferably in the abdomen for up to 4 weeks after the last dose of chemotherapy for a maximum of 26 weeks
  Interventions: Drug: Epoetin alfa 450 IU/kg once a week; Drug: Epoetin alfa 450 IU/kg once a week (QW)
- 002 (Experimental): Epoetin alfa 150 IU/kg 3 times a week (TIW) 150 IU/kg 3 times a week (TIW) by subcutaneous injection preferably in the abdomen for up to 4 weeks after the last dose of chemotherapy for a maximum of 26 weeks.
  Interventions: Drug: Epoetin alfa 150 IU/kg 3 times a week; Drug: Epoetin alfa 150 IU/kg 3 times a week (TIW)

INTERVENTIONS:
Drug: Epoetin alfa 450 IU/kg once a week — 450 IU/kg once a week by subcutaneous injection preferably in the abdomen for up to 4 weeks after the last dose of chemotherapy for a maximum of 26 weeks.
  Arms: 001
Drug: Epoetin alfa 150 IU/kg 3 times a week — 150 IU/kg 3 times a week by subcutaneous injection preferably in the abdomen for up to 4 weeks after the last dose of chemotherapy for a maximum of 26 weeks.
  Arms: 002
Drug: Epoetin alfa 450 IU/kg once a week (QW) — 450 IU/kg once a week (QW) by subcutaneous injection preferably in the abdomen for up to 4 weeks after the last dose of chemotherapy for a maximum of 26 weeks
  Arms: 001
Drug: Epoetin alfa 150 IU/kg 3 times a week (TIW) — 150 IU/kg 3 times a week (TIW) by subcutaneous injection preferably in the abdomen for up to 4 weeks after the last dose of chemotherapy for a maximum of 26 weeks.
  Arms: 002

SUMMARY:
The purpose of the study is to evaluate the safety of epoetin alfa in patients with cancer who have chemotherapy-related anemia.

DETAILED DESCRIPTION:
Epoetin alfa is an agent similar to a hormone produced in the kidney (ie, erythropoietin) that functions to increase the amount of red blood cells made in the bone marrow. This is a randomized (study drug assigned by chance), open-label (patients and their doctors will know the identity of study drug administered), safety study of 2 dosing regimens (doses and schedules) of epoetin alfa administered to patients with cancer who have chemotherapy-related anemia. Anemia is a lack of red blood cells that can result in symptoms of weakness, shortness of breath, fatigue, tiredness, and decreased activity. The primary outcome measure in the study is the number of patients in each treatment group with at least 1 clinically relevant and objectively confirmed (adjudicated) thrombovascular event (TVE) reviewed by an independent adjudication committee from Day 1 (baseline or the day of the first dose) through Week 16. An external review of relevant clinical data and medical imaging studies by an Adjudication Committee will be performed in a blinded fashion for confirmation of TVEs. The Adjudication Committee will confirm TVEs by reviewing all images (X-ray, Computed tomography [CT] scan, ultrasound, Magnetic Resonance Imaging [MRI] scan, etc) and other diagnostic procedures auch as coagulation tests or electrocardiograms in combination with a clinical patient profile as described for each specific type of TVE. Only TVEs that are determined by the Adjudication Committee to be clinically relevant and objectively confirmed will be counted in the analysis for the primary endpoint. Approximately 500 patients, who have cancer, are receiving chemotherapy, and are anemic, will take part in the study. Patients will participate in the study for up to 32 weeks (this includes a 2-week screening period to determine eligibility for the study, a 26-week treatment period, and a 4-week follow-up period to have end-of-study assessments [tests] performed). The length of participation in the study depends on the length of time the patient is receiving chemotherapy and epoetin alfa; patients in the study may receive up to a maximum of 26 weeks of treatment with epoetin alfa. Patients will be randomly assigned (assigned by chance like flipping a coin) to 1 of 2 treatment groups (Epoetin Alfa QW or Epoetin Alfa TIW). Patients assigned to the Epoetin Alfa QW Group will receive epoetin alfa at an initial dosage of 450 IU/kg once a week and patients assigned to Epoetin Alfa TIW Group will receive epoetin alfa 150 IU/kg 3 times a week by subcutaneous (underneath the skin) injection. Injections will be given preferably on Monday for patients in the Epoetin Alfa QW Group and on Mondays, Wednesdays, and Fridays for patients in the Epoetin Alfa TIW Group. During the study, patients will visit the study center weekly to have a blood sample collected to measure the amount of hemoglobin (red blood cells) in the blood. Depending on the hemoglobin level, the dose of epoetin alfa may be increased or decreased. Regardless of treatment group, if anemia does not improve in patients after 4 weeks of treatment, the dose of epoetin alfa will be increased to 300 IU/kg 3 times a week. If anemia does not improve after 4 weeks at the increased dose level of epoetin alfa (300 IU/kg 3 times a week), treatment with epoetin alfa will be stopped. In addition, during the study, patients may also receive treatment with iron supplements if the level of iron in the blood is low. During the study, safety will be monitored by evaluating adverse events and findings from clinical laboratory tests, 12-lead electrocardiograms (ECGs), blood pressure measurements, and physical examinations. Patients will receive epoetin alfa at an initial dose of 450 IU/kg once a week or 150 IU/kg 3 times a week by subcutaneous injection, preferably in the abdomen, for up to 4 weeks after the last dose of chemotherapy for a maximum of 26 weeks. Injections for Epoetin Alfa QW Group will be at the study center and for Epoetin TIW Group, the 1st weekly injection will be at the study center and the 2nd and 3rd weekly injections will be at the study center or at home by self-administration.

ELIGIBILITY:
Inclusion Criteria:

* Any nonmyeloid tumor confirmed by cytology and/or histology
* Day 1 baseline hemoglobin (Hb) level <=11 g/dL
* Expected to receive at least 12 weeks of chemotherapy after enrollment into the study
* Eastern Cooperative Oncology Group (ECOG) performance status <= 2

Exclusion Criteria:

* History of active second cancer except for adequately treated skin cancer and in situ (pre-invasive) cervical cancer
* History of deep venous thrombosis (DVT) (blood clots in the veins of the thighs or legs) or pulmonary embolism (PE) (blood clot in the lungs) within 12 months before study entry or at any time if the event is related to the current cancer, which is defined as diagnosis of the cancer within 3 months of a DVT/PE episode or a DVT/PE following the cancer diagnosis/treatment
* History of cardiovascular accident (CVA), transient ischemic attack (TIA) (stroke), acute coronary syndrome (ACS) (a condition indicating damage to the heart), or other arterial thrombosis (blood clots) within 6 months before study entry
* Onset of seizures within 3 months before randomization or poorly controlled seizures
* Brain tumor or brain metastasis from another malignancy or cardiac disease that is markedly or completely limiting, uncontrolled hypertension (high blood pressure), or anemia (a lack of red blood cells in the blood) for reasons other than cancer or chemotherapy
* Specifically excluded concomitant medications or therapies including prophylactic anticoagulation therapy for recurrence of prior thrombovascular event (TVE) (warfarin, unfractionated heparin, low molecular weight heparin [LMWH], except for prevention of central venous catheter thrombosis at doses specified in the protocol, direct thrombin inhibitors, or anti-platelet drugs [e.g., clopidogrel or ticlopidine]), except for prophylaxis in patients with known cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2006-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a randomized, open-label, multicenter study evaluating thrombovascular events in participants with cancer receiving chemotherapy and administered Epoetin Alfa once weekly (QW) or three times a week (TIW) for the treatment of anemia.
Groups:
- Epoetin Alfa QW: epoetin alfa at an initial dosage of 450 IU/kg once a week (QW)
- Epoetin Alfa TIW: epoetin alfa at an initial dosage of 150 IU/kg 3 times a week (TIW)
Period: Overall Study
Arm/Group | Epoetin Alfa QW | Epoetin Alfa TIW
Started | 242 | 262
Completed | 183 | 190
Not Completed | 59 | 72
Not completed — Adverse Event | 0 | 4
Not completed — Lack of Efficacy | 5 | 7
Not completed — Lost to Follow-up | 6 | 8
Not completed — Physician Decision | 1 | 3
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 20 | 17
Not completed — Chemotherapy Termination | 10 | 15
Not completed — Disease Progression | 7 | 7
Not completed — Prematurely Termination of Trial | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epoetin Alfa QW | Epoetin Alfa TIW | Total
Number analyzed (Participants) | 242 | 262 | 504
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 160 | 173 | 333
  >=65 years | 81 | 88 | 169
Age Continuous [Mean (Standard Deviation); unit: years] | 58.8 (13.35) | 57.5 (13.53) | 58.1 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156 | 181 | 337
  Male | 86 | 81 | 167
Region of Enrollment [Number; unit: participants]
  Bulgaria | 6 | 7 | 13
  France | 7 | 6 | 13
  Germany | 51 | 55 | 106
  Great Britain | 1 | 4 | 5
  Greece | 8 | 12 | 20
  Italy | 13 | 13 | 26
  Poland | 7 | 6 | 13
  Romania | 21 | 20 | 41
  Russia | 88 | 93 | 181
  Slovakia | 9 | 11 | 20
  Ukraine | 31 | 35 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least 1 Clinically Relevant and Objectively Confirmed Thrombovascular Event From Randomization Through Week 16
Description: Clinically relevant and objectively confirmed thrombovascular event (TVE) was determined by the Adjudication Committee from randomization through Week 16. Clinically relevant TVEs were defined as deep vein thrombosis (DVT) of the limbs; thromboses of other major veins; pulmonary embolism (PE);acute coronary syndrome (ACS);ischemic stroke of arterial or cardiac origin; cerebral venous thrombosis; and arterial thrombosis. Objectively confirmed was defined as the confirmation of the clinical diagnosis of a TVE by appropriate medical imaging studies and laboratory tests.
Time Frame: from randomization through Week 16
Population: The modified intent-to-treat (mITT) population was defined to include all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: particpants
Arm/Group | Epoetin Alfa QW | Epoetin Alfa TIW
Number analyzed (Participants) | 242 | 262
particpants | 5 | 10
Statistical Analysis 1: Comparison: Epoetin Alfa QW vs Epoetin Alfa TIW; The primary hypothesis was that the group of participants receiving epoetin alfa QW and the group of participants receiving epoetin alfa TIW would have similar incidence rate of participants with at least 1 clinically relevant and objectively confirmed TVE from randomization through Week 16; Test type: Superiority or Other; p = 0.248, Chi-squared; Risk Difference (RD) = -0.018, 95% CI 2-sided [-0.051 to 0.016]
Statistical Analysis 2: Comparison: Epoetin Alfa QW vs Epoetin Alfa TIW; Test type: Superiority or Other; p = 0.254, Regression, Logistic; Odds Ratio (OR) = 0.53, 95% CI [0.18 to 1.58]

2. Secondary Outcome: Number of Positively Adjudicated Thrombovascular Events
Description: The number of participants who have at least 1 clinically relevant and objectively confirmed (adjudicated) thrombovascular event (TVE) during the study.
Time Frame: during the study (randomization through week 26)
Population: The modified intent-to-treat (mITT) population used for safety analysis population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa QW | Epoetin Alfa TIW
Number analyzed (Participants) | 242 | 262
participants | 5 | 13
Statistical Analysis 1: Comparison: Epoetin Alfa QW vs Epoetin Alfa TIW; Test type: Superiority or Other; p = 0.08, Chi-squared; Risk Difference (RD) = -0.029, 95% CI 2-sided [-0.065 to 0.007]

3. Secondary Outcome: Time to First Positively Adjudicated Thrombovascular Event
Description: Analysis of time to first positively adjudicated thrombovascular event (TVE) measured from the date of randomization to the date of the first clinically relevant and objectively confirmed TVE as determined by the Adjudication Committee. Median time is non-estimable because of too few events, incidence was reported instead.
Time Frame: during the study (randomization through week 26)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa QW | Epoetin Alfa TIW
Number analyzed (Participants) | 242 | 262
participants | 5 | 13
Statistical Analysis 1: Comparison: Epoetin Alfa QW vs Epoetin Alfa TIW; Test type: Superiority or Other; p = 0.073, Log Rank; The stratified log-rank test accounting for ECOG performance status (0 or 1 versus 2) was used to compare the difference between treatment groups; Hazard Ratio (HR) = 0.40, 95% CI 2-sided [0.14 to 1.13] — The Cox regression model with covariates for treatment group and Eastern Cooperative Oncology Group (ECOG) performance status (0 or 1 versus 2) was used for estimates of hazard ratio and its 95% confidence interval

4. Secondary Outcome: Number of Suspected Thrombovascular Events
Description: Number of participants who have at least 1 suspected thrombovascular events (TVEs) during the entire study. Suspected TVEs were defined as suspected TVEs during the entire study, whether clinically relevant and objectively confirmed by the Adjudication Committee or not, whether confirmed by the investigator or not.
Time Frame: during the study (randomization through week 26)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa QW | Epoetin Alfa TIW
Number analyzed (Participants) | 242 | 262
participants | 9 | 20
Statistical Analysis 1: Comparison: Epoetin Alfa QW vs Epoetin Alfa TIW; Test type: Superiority or Other; p = 0.059, Chi-squared; Risk Difference (RD) = -0.039, 95% CI [-0.083 to 0.005]

5. Secondary Outcome: Time to First Suspected Thrombovascular Event
Description: Analysis of time to first suspected thrombovascular event (TVE) measured from the date of randomization to the date of the first suspected TVE during the study. Median time is non-estimable because of too few events, incidence was reported instead.
Time Frame: during the study (randomization through week 26)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa QW | Epoetin Alfa TIW
Number analyzed (Participants) | 242 | 262
participants | 9 | 20
Statistical Analysis 1: Comparison: Epoetin Alfa QW vs Epoetin Alfa TIW; Test type: Superiority or Other; p = 0.054, Log Rank; The stratified log-rank test accounting for ECOG score status (0 or 1 versus 2) was used to compare the difference between treatment groups; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.21 to 1.03] — The Cox regression model including covariates for treatment group and the Eastern Cooperative Oncology Group (ECOG) score status (0 or 1 versus 2) was used for estimates of a hazard ratio and its 95% confidence interval

6. Secondary Outcome: Mortality
Description: Number of participants who died during the study.
Time Frame: during the study (randomization through week 26)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa QW | Epoetin Alfa TIW
Number analyzed (Participants) | 242 | 262
participants | 25 | 26
Statistical Analysis 1: Comparison: Epoetin Alfa QW vs Epoetin Alfa TIW; Test type: Superiority or Other; p = 0.88, Chi-squared; Risk Difference (RD) = 0.0041, 95% CI [-0.0526 to 0.0608]

7. Secondary Outcome: Number of Hemoglobin Responders
Description: Hemoglobin response was defined as a hemoglobin increase of ≥2 g/dL from baseline or reaching a hemoglobin concentration of 12 g/dL, regardless of dose adjustment.
Time Frame: during the study (randomization through week 26)
Population: All participants who were randomized, regardless of whether or not they received study drug.
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa QW | Epoetin Alfa TIW
Number analyzed (Participants) | 242 | 262
participants | 179 | 187
Statistical Analysis 1: Comparison: Epoetin Alfa QW vs Epoetin Alfa TIW; Test type: Superiority or Other; p = 0.514, Chi-squared; Risk Difference (RD) = 0.026, 95% CI 2-sided [-0.056 to 0.108]

8. Secondary Outcome: Red Blood Cell Transfusions
Description: The number of participants who received at least 1 red blood cell (RBC) transfusion (packed RBC or whole blood) during the study.
Time Frame: during the study (randomization through week 26)
Population: All participants who were randomized, regardless of whether or not they received study drug.
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa QW | Epoetin Alfa TIW
Number analyzed (Participants) | 242 | 262
participants | 38 | 42
Statistical Analysis 1: Comparison: Epoetin Alfa QW vs Epoetin Alfa TIW; Test type: Superiority or Other; p = 0.920, Chi-squared; Risk Difference (RD) = -0.003, 95% CI 2-sided [-0.071 to 0.065]

ADVERSE EVENTS:
Arm/Group | Epoetin Alfa QW | Epoetin Alfa TIW
Serious Adverse Events (participants affected / at risk) | 53/242 | 64/262
Other Adverse Events (participants affected / at risk) | 157/242 | 151/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Alfa QW (N=242) | Epoetin Alfa TIW (N=262)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 | 20
Anaemia (Blood and lymphatic system disorders) | 4 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Pancytopenia (Blood and lymphatic system disorders) | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4
Pneumonia (Infections and infestations) | 2 | 9
Abscess jaw (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Erysipeloid (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 4
Hypotension (Vascular disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 2
Venous thrombosis limb (Vascular disorders) | 1 | 1
Cardiovascular insufficiency (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Subileus (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
General physical health deterioration (General disorders) | 2 | 1
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Chest pain (General disorders) | 0 | 2
Death (General disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Sudden cardiac death (General disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0
Pubic rami fracture (Injury, poisoning and procedural complications) | 0 | 1
Stent occlusion (Injury, poisoning and procedural complications) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Spinal cord compression (Nervous system disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 1
Aplasia (Congenital, familial and genetic disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Alfa QW (N=242) | Epoetin Alfa TIW (N=262)
Neutropenia (Blood and lymphatic system disorders) | 81 | 72
Thrombocytopenia (Blood and lymphatic system disorders) | 52 | 54
Leukopenia (Blood and lymphatic system disorders) | 51 | 44
Nausea (Gastrointestinal disorders) | 27 | 40
Diarrhoea (Gastrointestinal disorders) | 26 | 10
Vomiting (Gastrointestinal disorders) | 13 | 24
Asthenia (General disorders) | 21 | 14
Fatigue (General disorders) | 17 | 16
Pyrexia (General disorders) | 15 | 18
Anorexia (Metabolism and nutrition disorders) | 13 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the only disclosure restriction on the PI is that the sponsor has 60 days to review results communications prior to public release and can embargo communications regarding trial results for a period that does not exceed 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.